CLINICAL TRIAL: NCT05811351
Title: A Phase 2b, Randomized, Double-masked, Multicenter, Dose-ranging, Sham-controlled Clinical Trial to Evaluate Intravitreal JNJ-81201887 (AAVCAGsCD59) Compared to Sham Procedure for the Treatment of Geographic Atrophy (GA) Secondary to Age-related Macular Degeneration (AMD)
Brief Title: A Study to Evaluate Intravitreal JNJ-81201887 (AAVCAGsCD59) Compared to Sham Procedure for the Treatment of Geographic Atrophy (GA) Secondary to Age-related Macular Degeneration (AMD)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR109236; 81201887MDG2001 (Other: Janssen Research & Development, LLC); 2022-500746-16-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2023-03-07; First posted 2023-04-13 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Geographic Atrophy
Keywords: Macular Degeneration
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration | interventions — Prednisone; Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: JNJ-81201887 Low Dose (Experimental): Participants will receive a single low dose intravitreal injection of JNJ-81201887 in the study eye on Day 4. In addition, participants will receive a 20-day oral prednisone course starting on Day 1 and a single, long acting periocular triamcinolone (corticosteroid injection) on Day 4 for prophylaxis of intraocular inflammation.
  Interventions: Drug: JNJ-81201887; Drug: Prednisone; Drug: Triamcinolone
- Arm B: JNJ-81201887 High dose (Experimental): Participants will receive a single high dose intravitreal injection of JNJ-81201887 in the study eye on Day 4. In addition, participants will receive a 20-day oral prednisone course starting on Day 1 and a single, long acting periocular triamcinolone (corticosteroid injection) on Day 4 for prophylaxis of intraocular inflammation.
  Interventions: Drug: JNJ-81201887; Drug: Prednisone; Drug: Triamcinolone
- Arm C: Sham Procedure (Sham Comparator): Participants will receive sham procedure that matches the single JNJ21801887 injection on Day 4, a sham procedure that matches the long acting periocular triamcinolone (corticosteroid injection) on Day 4 and a 20-day placebo matching oral prednisone starting on Day 1.
  Interventions: Other: Placebo; Other: Sham Procedure

INTERVENTIONS:
Drug: JNJ-81201887 — JNJ-81201887 will be administered as intravitreal injection.
  Other Names: AAVCAGsCD59
  Arms: Arm A: JNJ-81201887 Low Dose; Arm B: JNJ-81201887 High dose
Drug: Prednisone — Prednisone will be administered as oral capsule.
  Arms: Arm A: JNJ-81201887 Low Dose; Arm B: JNJ-81201887 High dose
Other: Placebo — Prednisone matching placebo will be administered as oral capsule.
  Arms: Arm C: Sham Procedure
Drug: Triamcinolone — Triamcinolone (corticosteroid injection) periocular injection will be administered as per local practice.
  Arms: Arm A: JNJ-81201887 Low Dose; Arm B: JNJ-81201887 High dose
Other: Sham Procedure — Sham injections matching to single JNJ-81201887 injection and matching to corticosteroid (triamcinolone) periocular injection will be administered.
  Arms: Arm C: Sham Procedure

SUMMARY:
The purpose of this study is to evaluate change in geographic atrophy (GA) lesion growth of eyes treated with JNJ-81201887 compared to sham control.

ELIGIBILITY:
Inclusion Criteria:

* Have non-subfoveal (defined as not involving the center point of the fovea) geographic atrophy (GA) secondary to age-related macular degeneration (AMD) with an area that can be measured and measures 2.5 millimeter square (mm^2) to 17.5 mm^2 (1- and 7- disc areas respectively), determined by the central reading center (CRC) from screening images of fundus autofluorescence (FAF) and spectral domain optical coherence tomography (SD-OCT)
* If GA is multifocal, at least one focal lesion must be greater than or equal to (>=) 1.25 mm^2 (0.5- disc area), as assessed by the CRC
* GA can be photographed in its entirety by FAF, using a 30- degree image centered on the fovea, as assessed by the CRC
* Fellow eye must be present with a best corrected distance visual acuity (BCVA) of counting fingers or better
* Man or woman (according to their reproductive organs and functions assigned by chromosomal complement)

Exclusion Criteria:

* History of transpupillary thermotherapy, photodynamic therapy or external-beam radiation therapy in the region of study eye
* Any prior thermal laser in the macular region, regardless of indication
* History of retinal detachment (with or without repair)
* Active, infectious conjunctivitis, keratitis, scleritis, or endophthalmitis
* Any sign of diabetic retinopathy or central serous chorioretinopathy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2026-02-26 (Estimated); Study Completion 2026-02-26 (Estimated)

PRIMARY OUTCOMES:
Global: Change From Baseline in Square Root of Geographic Atrophy (GA) Lesion Area in the Study Eye at Month 18 | Baseline and Month 18
  Change from baseline in GA lesion area in the study at month 18 eye will be measured via retinal imaging using fundus auto fluorescence (FAF).
United States (U.S.) Specific: Rate of Change in Untransformed GA Lesion Area in the Study Eye | Baseline to Month 18
  Rate of Change in untransformed GA lesion area in the study eye will be measured via retinal imaging using FAF. A piecewise linear mixed effects (PLME) model will be used for the primary efficacy analysis for rate of change in GA area (GAA) in the study eye.

SECONDARY OUTCOMES:
Change From Baseline in Low Luminance Visual Acuity (LLVA) at Month 18 | Baseline and Month 18
  Best corrected LLVA will be assessed using the early treatment diabetic retinopathy study (ETDRS) chart at a starting distance of 4 meter.
Change From Baseline in Reading Speed at Month 18 | Baseline and Month 18
  Change from baseline in reading speed (normal luminance) as assessed by Radner reading charts will be performed in the study eye and binocularly for participants who are fluent in the languages available for the Radner Chart will be reported.
Change From Baseline in Retinal Sensitivity by Mesopic Microperimetry (MAIA) at Month 18 | Baseline and Month 18
  Change from baseline retinal sensitivity by MAIA will be reported.
Change From Baseline in Best Corrected Visual Acuity (BCVA) at Month 18 | Baseline and Month 18
  Change from baseline in BCVA will be reported and this will be measured using the ETDRS chart at a starting distance of 4 meter.
Change From Baseline in Functional Reading Independence (FRI) Index at Month 18 | Baseline and Month 18
  The FRI is an interviewer-administered questionnaire with 7 items on functional reading activities most relevant to GA AMD participants. Item scores reflect decreasing levels of functional reading independence. The FRI Index yields continuous mean scores (range 1 to 4), and ordinal-level scores from Level 1 = "Unable to do" to Level 4 = "Totally independent." For each FRI Index reading activity performed in the past 7 days, participants are asked about the extent to which they required vision aids, adjustments in the activity, or help from another person.
Change From Baseline in National Eye Institute Visual Functioning Questionnaire-25 (NEI-VFQ-25) Composite Score at Month 18 | Baseline and Month 18
  The 2000 version of the NEI-VFQ-25, which must be interviewer-administered, includes 25 items and is scored to produce 11 subscales and a general health item. The 11 subscales include General Vision (1 item), Ocular Pain (2 items), Near Activities (3 items), Distance Activities (3 items), Social Functioning (2 items), Mental Health (2 items), Role Difficulties (2 items), Dependency (3 items), Driving (3 items), Color Vision (1 item), and Peripheral Vision (1 item). Response to each question converted to 0-100 score. Each subscale, total score equal to (=) average of items contributing to score. For each subscale and total score, score range: 0 to 100, higher score equal to less symptoms/better visual functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (162):
- United States (79):
  - Retinal Research Institute, Phoenix, Arizona
  - Retina Associates Southwest PC, Tucson, Arizona
  - Retina Consultants of Orange County, Fullerton, California
  - Retina Associates Of Southern California, Huntington Beach, California
  - Shiley Eye Institute Jacobs Retina Center, La Jolla, California
  - Jules Stein Eye Institute UCLA, Los Angeles, California
  - The Retina Partners, Los Angeles, California
  - California Retina Consultants, Oxnard, California
  - Stanford Health Care, Palo Alto, California
  - California Eye Medical Specialists, Pasadena, California
  - Retina Consultants San Diego, Poway, California
  - Retina Consultants of Southern California, Redlands, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Colorado Retina - Lakewood Clinic, Lakewood, Colorado
  - Retina Group of Florida, Fort Lauderdale, Florida
  - National Opthalmic Research Institute, Fort Myers, Florida
  - VitreoRetinal Associates, PA, Gainesville, Florida
  - MedEye Associates, Miami, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - East Florida Eye Institute, Stuart, Florida
  - Georgia Retina, Marietta, Georgia
  - Marietta Eye Clinic, Marietta, Georgia
  - University Of Illinois, Chicago, Illinois
  - Retina Associates, Elmhurst, Illinois
  - University Retina, Lemont, Illinois
  - Midwest Eye Institute, Carmel, Indiana
  - Maine Eye Center, Portland, Maine
  - Retina Specialists, Baltimore, Maryland
  - The Retina Care Center, Baltimore, Maryland
  - The Retina Group of Washington, Chevy Chase, Maryland
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Vitreo Retinal Associates-Worcester, Worcester, Massachusetts
  - Foundation for Vision Research, Grand Rapids, Michigan
  - Associated Retinal Consultants P.C., Royal Oak, Michigan
  - Retina Consultants of Minnesota, Saint Louis Park, Minnesota
  - The Retina Institute, St Louis, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - Wills Eye/Mid Atlantic Retina, Cherry Hill, New Jersey
  - Long Island Vitreo Retinal Consultants, Great Neck, New York
  - Retina-Vitreous Surgeons of Central New York, Liverpool, New York
  - Vitreous Retina Macula Consultants of New York, New York, New York
  - Retina Consultants PLLC, Slingerlands, New York
  - Opthalmic Consultants of the Capital Region, Troy, New York
  - Asheville Eye Associates - Western Carolina Retinal Associates, Asheville, North Carolina
  - Duke University, Durham, North Carolina
  - Graystone Eye, Hickory, North Carolina
  - NC Retina Associates, Wake Forest, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Verum Research LLC, Eugene, Oregon
  - Casey Eye Institute, Portland, Oregon
  - Cascade Medical Research Institute, LLC, Springfield, Oregon
  - Erie Retina Research, Erie, Pennsylvania
  - Charleston Neuroscience Institute, LLC, Beaufort, South Carolina
  - Charles Retina Institute, Germantown, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Panhandle Eye Group LLP-Southwest Retina Specialists, Amarillo, Texas
  - Austin Clinical Research, Austin, Texas
  - Retina and Vitreous of Texas, PLLC, Bellaire, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Retina Foundation of the Southwest, Dallas, Texas
  - Texas Retina Associates, Dallas, Texas
  - UT Southwestern, Dallas, Texas
  - Texas Retina Associates, Fort Worth, Texas
  - Houston Eye Associates, Houston, Texas
  - San Antonio Eye Center, San Antonio, Texas
  - Retina Associates Of South Texas P A, San Antonio, Texas
  - Retina Consultants of Texas, San Antonio, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
  - Strategic Clinical Research Group, Willow Park, Texas
  - Retina Associates of Utah P C, Salt Lake City, Utah
  - Rocky Mountain Retina Consultants, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah
  - Piedmont Eye Center, Lynchburg, Virginia
  - Wagner Kapoor Research institute, Norfolk, Virginia
  - Spokane Eye Clinical Research, Spokane, Washington
- Australia (5):
  - Adelaide Eye and Retina Centre, Adelaide
  - Centre for Eye Research Australia, East Melbourne
  - Strathfield Retina Clinic, Strathfield
  - Sydney Retina Clinic and Day Surgery, Sydney
  - Sydney West Retina, Westmead
- Belgium (4):
  - Ziekenhuis Oost-Limburg, Genk
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire de Liege Domaine Universitaire du Sart Tilman, Liège
- Canada (5):
  - Calgary Retina Consultants, Calgary, Alberta
  - Alberta Retina Consultants, Edmonton, Alberta
  - The Ottawa Hospital Research Institute, Ottawa, Ontario
  - The Retina Centre of Ottawa, Ottawa, Ontario
  - Institut De L'oeil Des Laurentides, Boisbriand, Quebec
- Czechia (3):
  - OFTEX Ltd. - EYE CENTER, Pardubice
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - AXON Clinical s.r.o., Prague
- Denmark (3):
  - Aalborg University Hospital, Aalborg
  - University Hospital Of Copenhagen, Glostrup Hospital, Glostrup Municipality
  - Zealand University Hospital, Roskilde
- Germany (11):
  - Charite Universitaetsmedizin Berlin, Berlin
  - Universitaets-Augenklinik Bonn, Bonn
  - Universitatsklinikum Gießen - Klinik und Poliklinik fur Augenheilkunde, Giessen
  - Klinikum Gottingen der Georg August Universitat, Göttingen
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinikum Schleswig Holstein Kiel, Kiel
  - Universitaetsklinikum Leipzig, Leipzig
  - Klinikum Ludwigshafen, Ludwigshafen am Rhein
  - Augenzentrum am St Franziskus Hospital Munster, Münster
  - Universitaetsklinikum Muenster, Münster
  - Universitaetsklinikum Tuebingen, Tübingen
- Hungary (3):
  - Eszak Pesti Centrumkorhaz Honvedkorhaz, Budapest
  - Ganglion Orvosi Központ, Pécs
  - Zala Megyei Szent Rafael Korhaz, Zalaegerszeg
- Italy (6):
  - Arcispedale S. Anna Ferrara, Ferrara
  - Fondazione IRCCS Ca Granda Ospedale Policlinico Di Milano, Milan
  - Ospedale San Raffaele, Milan
  - Sacco Hospital, Milan
  - Azienda Ospedaliera Univ.- Università Degli studi della Campania - Luigi Vanvitelli, Napoli
  - Policlinico Universitario Agostino Gemelli, Roma
- Netherlands (3):
  - Amsterdam University Medical Centers Location Academic Medical Center, Amsterdam
  - Radboudumc, Nijmegen
  - Het Oogziekenhuis Rotterdam, Rotterdam
- Poland (4):
  - Oculomedica, Bydgoszcz
  - Oftalmika, Bydgoszcz
  - Uno Med, Tarnów
  - Warszawski Szpital Okulistyczny, Warsaw
- Portugal (3):
  - Uls Coimbra - Hosp. Univ. Coimbra, Coimbra
  - Espaco Medico de Coimbra, Coimbra
  - Uls Sao Joao - Hosp. Sao Joao, Porto
- Spain (18):
  - Centro de Oftalmologia Barraquer, Barcelona
  - Centro Medico Teknon S.L., Barcelona
  - Inst. Cat. de Retina, Barcelona
  - Hosp. Dos de Maig, Barcelona
  - Inst. de Microcirugia Ocular, Barcelona
  - Clinica Oftalvist Valencia, Burjassot
  - Hosp. La Arruzafa, Córdoba
  - Hosp. Univ. Donostia, Donostia / San Sebastian
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Clinica Baviera Madrid Castellana, Madrid
  - Hosp. Univ. Pta. de Hierro Majadahonda, Majadahonda
  - Clinica Univ. de Navarra, Pamplona
  - Idc Salud Hosp. Gral. de Catalunya, Sant Cugat del Vallès
  - Hosp. Prov. Do Conxo, Santiago de Compostela
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Clinico Univ. Lozano Blesa, Zaragoza
  - Hosp. Univ. Miguel Servet, Zaragoza
- S:t Eriks Ogonsjukhus, Stockholm, Sweden
- Inselspital Universitatsspital Bern, Bern, Switzerland
- Turkey (Türkiye) (5):
  - Hacettepe University Hospital, Ankara
  - Baskent University Ankara Hospital, Ankara
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Dokuz Eylul University Hospital, Izmir
  - Konya Selcuk University Medical Faculty, Konya
- United Kingdom (8):
  - Bristol Eye Hospital, Bristol
  - Moorfields Eye Hospital, London
  - Central Middlesex Hospital, London
  - The Retina Clinic London, London
  - Manchester Royal Eye Hospital, Manchester
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Oxford Eye Hospital, Oxford
  - Southampton University Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency